CLINICAL TRIAL: NCT00706394
Title: Prospective, Multicenter, Single Arm Phase II Study of the Powerlink 34mm Cuff for the Endovascular Repair of Abdominal Aortic Aneurysms
Brief Title: 34mm Cuff Study for Endovascular Repair of Abdominal Aortic Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP03-023
Record Dates: First submitted 2008-05-02; First posted 2008-06-27 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Powerlink; 34mm; Abdominal Aortic Aneurysm; EVAR
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Powerlink 34mm cuff stent graft
  Interventions: Device: Endologix Powerlink 34 mm stent graft cuff

INTERVENTIONS:
Device: Endologix Powerlink 34 mm stent graft cuff — Endovascular abdominal aortic aneurysm repair
  Other Names: Endologix Powerlink 34mm cuff [model 34-34-80L]

SUMMARY:
Study of anatomical fixation with a 34mm proximal extension

DETAILED DESCRIPTION:
The 34mm proximal extension stent graft is intended to augment the primary 28mm infrarenal bifurcated stent graft to accommodate patient anatomy (neck diameters up to 32mm) and provide an effective seal to prevent/repair proximal Type I endoleaks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Informed consent understood and signed
* Will comply with protocol follow-up requirements
* Candidate for conventional open surgical repair
* Aneurysm outer diameter is one or more of the following:

  * greater than or equal to 4.0cm
  * greater than or equal to 3.0cm (saccular aneurysm)
  * greater than or equal to twice the normal aortic outer diameter
  * rapidly growing (greater than or equal to 5mm over 6 months)
* Proximal non-aneurysmal aortic neck fixation length greater than or equal to 1.5cm between the renal arteries and the aneurysm
* Non-aneurysmal proximal aortic neck inner diameter between 23 and 32mm
* Iliac artery internal diameter greater than or equal to 8 mm

Exclusion Criteria:

* Life expectancy <2 years
* Participating in another clinical study
* Pregnant or lactating women
* Acutely ruptured/leaking aneurysm
* Traumatic vascular injury
* Other medical or psychiatric problems
* Contraindication to non-ionic contrast media or anticoagulants
* Coagulopathy or bleeding disorder
* Active systemic or localized groin infection
* Indispensable inferior mesenteric artery
* Connective tissue disease (e.g., Marfan's Syndrome)
* Creatinine level >1.7 mg/dl
* Renal transplant patient
* Proximal attachment site >60º angle to the aneurysm body
* Iliac arteries >90º angle
* <1.5 cm of non-aneurysmal common iliac artery above the iliac bifurcation on both sides [One internal iliac artery is required to remain patent]
* Thrombus >30% at implantation site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-08-10 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Y Woo, MD, Principal Investigator — Hospital at the University of Pennsylvania, Philadelphia, PA 19104, United States; O. W. Brown, MD, Principal Investigator — William Beaumont Hospital, Royal Oak, MI 48073, United States; James G. Melton, DO, Principal Investigator — Oklahoma Cardiovascular Research Group, Oklahoma City, OK 73120, United States; Steven H. Tyndall, MD, Principal Investigator — Nebraska Heart Hospital, Lincoln, NE 68526, United States; William M. Moore, MD, Principal Investigator — Lexington Medical Center, West Columbia, SC 29169, United States; Salem George, MD, Principal Investigator — Baptist Hospital East, Louisville, KY 40207, United States; Kerry C. Prewitt, MD, Principal Investigator — St. Joseph Medical Center, Towson, MD 21204, United States; Paul Anain, MD, Principal Investigator — Sisters of Charity Hospital, Buffalo, NY 14214, United States; Robert Beasley, MD, Principal Investigator — Mount Sinai Medical Center, Miami Beach, FL 33140, United States; Barry T. Katzen, MD, Principal Investigator — Baptist Cardiac and Vascular Institute, Miami, FL 33176, United States
Locations (10):
- United States (10):
  - Mount Sinai Medical Center, Miami, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Baptist Hospital East, Louisville, Kentucky
  - St. Joseph Medical Center, Towson, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Sisters of Charity Hospital, Buffalo, New York
  - Oklahoma Cardiovascular Associates, Oklahoma City, Oklahoma
  - Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Lexington Medical Center, West Columbia, South Carolina

REFERENCES:
- [Result] Jordan WD Jr, Moore WM Jr, Melton JG, Brown OW, Carpenter JP; Endologix Investigators. Secure fixation following EVAR with the Powerlink XL System in wide aortic necks: results of a prospective, multicenter trial. J Vasc Surg. 2009 Nov;50(5):979-86. doi: 10.1016/j.jvs.2009.05.057. Epub 2009 Aug 12. PMID 19679425

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy: Powerlink 34mm cuff stent graft
  Endologix Powerlink 34 mm stent graft cuff: Endovascular abdominal aortic aneurysm repair
Period: Overall Study
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Started | 19
Completed | 8
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: All participants received a commercially available 28mm Powerlink infrarenal bifurcated stent graft and a 34mm infrarental proximal cuff
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Medical History [Count of Participants; unit: Participants]
  Angina | 2
  Arrhythmia | 6
  Cancer | 4
  Cerebrovascular Disease | 6
  Coagulopathy | 1
  Congestive Heart Failure | 3
  Coronary artery Disease | 10
  COPD | 11
  Diabetes | 3
  Family History of AAA | 3
  Gastrointestinal abnormality | 7
  Hypertension | 17
  Hypercholesterolemia | 14
  Liver Disease | 0
  Peripheral Occlusive Arterial Disease | 9
  Prior Abdominal Surgery | 7
  Prio MI (>6 mo) | 1
  Prio MI (< 6 mo) | 0
  CABG | 3
  PTCA/Stent | 4
  Renal Failure | 1
  Smoking (ever) | 19
  Valvular Disease | 2
  Valve Replacement | 1
Aneurysm Diameter Distribution [Count of Participants; unit: Participants]
  <30mm | 0
  30mm to 39mm | 0
  40mm to 49mm | 2
  50mm to 59mm | 14
  60mm to 69mm | 2
  70mm to 79mm | 0
  >79mm | 1
Mean Aneurysm Measurements [Mean (Standard Deviation); unit: mm]
  External Iliac Diameter | 9.3 (1.2)
  Proximal non-aneurysmal neck diameter | 28 (1.9)
  Distal non-aneurysmal neck diameter | 31 (1.4)
  Maximum Aneurysm Diameter | 57 (12)
  Proximal non-aneurysmal right iliac diameter | 15 (2.7)
  Distal non-aneurysmal right iliac diameter | 13 (2.3)
  Proximal non-aneurysmal left iliac diameter | 15 (3.4)
  Distall non-aneurysmal left iliac diameter | 13 (2.6)
  Proximal Seal Zone lenght | 27 (11)
  Length Proximal Neck to Left Proximal Iliac | 122 (21)
  Length Proximal Neck to Distal Right Iliac | 171 (23)
  Length Proximal Neck to Distal Left Iliac | 169 (23)
  Right Distal Seal Zone Length | 41 (13)
  Left Distal Seal Zone Length | 38 (13)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Proximal Type I Endoleak at Each Timepoint
Description: Percentage of patients with Type Ia endoleaks at each timepoint (discharge, 1, 6, 12, 24, 36, 48 and 60 months).
Time Frame: Five years
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy: Powerlink 34mm cuff stent graft
  Endologix Powerlink 34 mm stent graft cuff used for Endovascular abdominal aortic aneurysm repair
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Participants
  Discharge | 1
  1 Month | 0
  6 Months | 0
  12 Months | 0
  24 Months | 0
  48 Months | 0
  60 Months | 0

2. Secondary Outcome: Number of Participants With Successful Delivery and Deployment of the Device
Description: Successful delivery and deployment of the device with no complication.
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Participants | 19

3. Secondary Outcome: Number of Participants With Type III Endoleaks at Each Timepoint
Description: Percentage of patients with a Type III endoleaks at the timepoints (1, 6, 12, 24, 36, 48 and 60 Months) as reported by CoreLab.
Time Frame: 5 Years
Population: Results are provided as the number of events over the number of patients with the follow-up image available.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Participants
  1 Month: number analyzed (Participants) | 16
  1 Month | 0
  6 Months: number analyzed (Participants) | 14
  6 Months | 0
  12 Months: number analyzed (Participants) | 12
  12 Months | 0
  24 Months: number analyzed (Participants) | 14
  24 Months | 0
  36 Months: number analyzed (Participants) | 9
  36 Months | 0
  48 Months: number analyzed (Participants) | 7
  48 Months | 0
  60 Months: number analyzed (Participants) | 6
  60 Months | 0

4. Secondary Outcome: Number of Participants With Stent Fracture at Each Timepoint
Description: Percentage of patients with a stent fracture over the timepoints (1, 6, 12, 24, 36, 48 and 60 Months) as reported by the CoreLab.
Time Frame: 5 Years
Population: Results are provided as the number of events over the number of patients with the follow-up image available.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Participants
  Discharge: number analyzed (Participants) | 12
  Discharge | 0
  1 Month: number analyzed (Participants) | 18
  1 Month | 0
  6 Months: number analyzed (Participants) | 16
  6 Months | 0
  12 Months: number analyzed (Participants) | 12
  12 Months | 0
  24 Months: number analyzed (Participants) | 16
  24 Months | 0
  36 Months: number analyzed (Participants) | 9
  36 Months | 0
  48 Months: number analyzed (Participants) | 7
  48 Months | 0
  60 Months: number analyzed (Participants) | 6
  60 Months | 0

5. Secondary Outcome: Number of Participants With Stent Graft Obstruction at Each Timepoint
Description: Percentage of patients with a stent graft obstruction at each timepoint (1, 6, 12, 24, 36, 48 and 60 Months) as reported by Corelab.
Time Frame: 5 Years
Population: Results are provided as the number of events over the number of patients with the follow-up image available.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Participants
  1 Month: number analyzed (Participants) | 16
  1 Month | 0
  6 Months: number analyzed (Participants) | 14
  6 Months | 0
  12 Months: number analyzed (Participants) | 12
  12 Months | 0
  24 Months: number analyzed (Participants) | 13
  24 Months | 0
  36 Months: number analyzed (Participants) | 9
  36 Months | 0
  48 Months: number analyzed (Participants) | 6
  48 Months | 0
  60 Months: number analyzed (Participants) | 6
  60 Months | 0

6. Secondary Outcome: Number of Participants With Migration at Each Timepoint
Description: Percentage of patients presenting a migration at each timepoint (1, 6, 12, 24, 36, 48, 60 Months) as reported by Corelab.
Time Frame: 5 Years
Population: Results are provided as the number of events over the number of patients with the follow-up image available.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Participants
  1 Month: number analyzed (Participants) | 16
  1 Month | 0
  6 Months: number analyzed (Participants) | 14
  6 Months | 0
  12 Months: number analyzed (Participants) | 12
  12 Months | 0
  24 Months: number analyzed (Participants) | 13
  24 Months | 0
  36 Months: number analyzed (Participants) | 9
  36 Months | 0
  48 Months: number analyzed (Participants) | 6
  48 Months | 0
  60 Months: number analyzed (Participants) | 6
  60 Months | 0

7. Secondary Outcome: Number of Participants With Type II Endoleaks at Each Timepoint
Description: Percentage of patients with Type II endoleak at each time point (1, 6, 12, 24, 36, 48 and 60 Months) as reported by CoreLab.
Time Frame: 5 Years
Population: Results are provided as the number of events over the number of patients with the follow-up image available.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Participants
  1 Month: number analyzed (Participants) | 16
  1 Month | 4
  6 Months: number analyzed (Participants) | 14
  6 Months | 2
  12 Months: number analyzed (Participants) | 12
  12 Months | 0
  24 Months: number analyzed (Participants) | 14
  24 Months | 2
  36 Months: number analyzed (Participants) | 9
  36 Months | 1
  48 Months: number analyzed (Participants) | 7
  48 Months | 1
  60 Months: number analyzed (Participants) | 6
  60 Months | 0

8. Secondary Outcome: Number of Participants With Aneurysm Diameter Change at Each Timepoint
Description: Percentage of patients with a decrease, stable or increase aneurysm diameter at 6, 12, 24, 36, 48 and 60 Months compared to 1 Month as reported by CoreLab.
Time Frame: 5 Years
Population: Results are provided as the number of events over the number of patients with the follow-up image available.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
Participants
  6 Months: number analyzed (Participants) | 14
  6 Months: Decrease | 3
  6 Months: Stable | 11
  6 Months: Increase | 0
  12 Months: number analyzed (Participants) | 12
  12 Months: Decrease | 3
  12 Months: Stable | 9
  12 Months: Increase | 0
  24 Months: number analyzed (Participants) | 16
  24 Months: Decrease | 6
  24 Months: Stable | 10
  24 Months: Increase | 0
  36 Months: number analyzed (Participants) | 9
  36 Months: Decrease | 6
  36 Months: Stable | 3
  36 Months: Increase | 0
  48 Months: number analyzed (Participants) | 7
  48 Months: Decrease | 4
  48 Months: Stable | 3
  48 Months: Increase | 0
  60 Months: number analyzed (Participants) | 6
  60 Months: Decrease | 3
  60 Months: Stable | 2
  60 Months: Increase | 1

9. Secondary Outcome: Maximum Diameter Measurements
Description: Maximum Diameter changes compared to the pre-operative at each timepoint (1, 6, 12, 24, 36, 48 Months).
Time Frame: 5 Years
Population: Results are provided as the number of events over the number of patients with the follow-up image available.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
mm
  Pre-operative: number analyzed (Participants) | 16
  Pre-operative | 56 (15)
  1 Month: number analyzed (Participants) | 16
  1 Month | 57 (15)
  6 Months: number analyzed (Participants) | 14
  6 Months | 56 (16)
  12 Months: number analyzed (Participants) | 12
  12 Months | 56 (18)
  24 Months: number analyzed (Participants) | 14
  24 Months | 52 (17)
  36 Months: number analyzed (Participants) | 9
  36 Months | 46 (8)
  48 Months: number analyzed (Participants) | 7
  48 Months | 45.5 (9)
  60 Months: number analyzed (Participants) | 6
  60 Months | 47.3 (13)

10. Secondary Outcome: Aneurysm Volume Measurements
Description: Aneurysm Volume changes over each time point (1, 6, 12, 24, 36, 48 and 60 Months) compared to pre-operative as reported by CoreLab.
Time Frame: 5 Years
Population: Results are provided as the number of events over the number of patients with the follow-up image available.
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Single Arm 34mm Infrarenal Cuff for Treatment of Patients With Larger Aortic Neck Anatomy
Number analyzed (Participants) | 19
cm3
  Pre-operative: number analyzed (Participants) | 16
  Pre-operative | 203 (125)
  1 Month: number analyzed (Participants) | 16
  1 Month | 213 (136)
  6 Months: number analyzed (Participants) | 14
  6 Months | 217 (136)
  12 Months: number analyzed (Participants) | 12
  12 Months | 213 (136)
  24 Months: number analyzed (Participants) | 14
  24 Months | 164 (49)
  36 Months: number analyzed (Participants) | 9
  36 Months | 163 (51)
  48 Months: number analyzed (Participants) | 7
  48 Months | 166 (60)
  60 Months: number analyzed (Participants) | 6
  60 Months | 161 (47)

ADVERSE EVENTS:
Time Frame: Up to 5 Years
Groups:
- Powerlink 34mm Cuff Stent Graft: Powerlink 34mm cuff stent graft
  Endologix Powerlink 34 mm stent graft cuff used for Endovascular abdominal aortic aneurysm repair
Arm/Group | Powerlink 34mm Cuff Stent Graft
All-Cause Mortality (participants affected / at risk) | 6/19
Serious Adverse Events (participants affected / at risk) | 14/19
Other Adverse Events (participants affected / at risk) | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Powerlink 34mm Cuff Stent Graft (N=19)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Decreased Hematocrit (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
MI (Cardiac disorders) | 1 (1)
Triple Vessel Coronary Artery Disease (Cardiac disorders) | 1 (1)
Cholecystis (Gastrointestinal disorders) | 1 (1)
Erosive Gastritis/Epgastric Pain (Gastrointestinal disorders) | 1 (1)
GI Bleeding (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Vomiting, Diarrhea, Dehydration (Gastrointestinal disorders) | 1 (1)
Increased Ascites secondary to cirrhosis (Gastrointestinal disorders) | 1 (1)
Lieus (Gastrointestinal disorders) | 1 (1)
Pseudomembraneous colitis (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Non cardiac CP (General disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (2)
Left groin incision infection (Infections and infestations) | 1 (1)
MRSA left lower leg (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Compression Fracture of Lumbar Spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Umbilical Hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Brain Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic Brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Side branch-type pancreatic papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Stage IV small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Left lower lung mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endoleak with Increased aneurysm (Product Issues) | 1 (1)
Limb extension right distal leak (Product Issues) | 1 (1)
Type I endoleak requiring endovascular repair (Product Issues) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Major depression recurrent (Psychiatric disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right leg ulcer and tingling (Skin and subcutaneous tissue disorders) | 1 (1)
Translumbar embolization of AAA sac (Surgical and medical procedures) | 1 (1)
Aneurysm increased >/=5mm (Vascular disorders) | 1 (1)
Coagulopathy: decreased platelets due to HIT+ (Vascular disorders) | 1 (1)
Ischemic Left Leg (Vascular disorders) | 1 (1)
Left femoral-popliteal bypass with graft (Vascular disorders) | 1 (1)
Right femoral tibial bypass for gangrenous foot (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Powerlink 34mm Cuff Stent Graft (N=19)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Vision problems (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Postop ileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Peri rectal abscess (Gastrointestinal disorders) | 1 (1)
Burning down left anterior leg (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Mild erythema left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Right inguinal hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Endoleak Type I distal (Product Issues) | 1 (1)
Endoleak Type II IMA (Product Issues) | 1 (1)
Left distal endoleak (Product Issues) | 1 (1)
Type I endoleak (Product Issues) | 1 (1)
Type I endoleak - placement aortic stent (Product Issues) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion postop (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Severe Pulmonary Enphisema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ABO Sugical Incisional Pain (Surgical and medical procedures) | 1 (1)
Incisional pain (Surgical and medical procedures) | 1 (1)
Left groin bleed (Surgical and medical procedures) | 1 (1)
Removal of sternal wire - non healing (Surgical and medical procedures) | 1 (1)
Carotid endoarterectomy (Vascular disorders) | 1 (1)
Carotid Stenosis (Vascular disorders) | 1 (1)
Elevated velocity left internal carotid (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Renal Artery stenosis (Vascular disorders) | 1 (1)
Increased Creatinine (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less